CLINICAL TRIAL: NCT05496127
Title: Two Different Approaches in Patients With Chronic Neck Pain: Sensorimotor Exercises Practice and Yoga
Brief Title: Sensorimotor Exercises Practice and Yoga in Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Dilanur Özkaraoğlu, PT, MSc, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-34229
Record Dates: First submitted 2022-07-19; First posted 2022-08-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain; Neck Pain
MeSH Terms: conditions — Chronic Pain; Neck Pain | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor Exercise Group (Experimental): Sensorimotor exercise group; oculomotor exercise to provide information from the visual system, laser target exercise to provide information from the proprioception system, and postural stability exercise to provide information from the vestibular system. Within the scope of oculomotor exercise, gaze stability exercise and head-body coordination exercise will be given to the participants. Laser target exercise will be given with the laser target fixed on the participant's head and 90 cm away from the target. Postural stability exercise will be given in the form of tandem exercise and standing on one leg.
  Interventions: Other: Sensorimotor Exercises and Yoga
- Yoga Exercise Group (Experimental): Yoga group will be given yoga exercises including 14 poses. These exercises are: bridge pose, corpse pose, bharadvaja's twist, downward facing dog, downward facing hero, extended side angle, extended triangle, mountain pose, prosperous pose, reclining big toe, standing half forward bend, thunderbolt pose, upward hand pose, warrior pose II.
  Interventions: Other: Sensorimotor Exercises and Yoga

INTERVENTIONS:
Other: Sensorimotor Exercises and Yoga — Within the content of sensorimotor exercise; oculomotor exercise, laser target exercise and postural stability exercise were applied. 14 yoga poses were applied within the content of Yoga Exercises.

SUMMARY:
Neck pain is an important public health problem with a high lifetime prevalence and frequently occurring in all industrialized countries. Clinical practice guidelines for chronic neck pain recommend conservative management. Conservative treatment includes many approaches such as endurance, stretching and strengthening exercises, manual therapy, proprioceptive exercises, pilates and yoga. In patients with chronic neck pain, atrophy of deep neck muscles, deterioration in fiber type ratio, muscle tenderness and decreased range of motion are observed. These problems cause poor cervical postural control system and thus impaired sense of proprioception, loss of balance, decreased eye movement and cervical muscle activity. Sensorimotor control of upright posture and head-eye movement relies on information from the vestibular, visual, and proprioceptive systems that assemble throughout the central nervous system.The cervical spine has an important role in providing proprioceptive input. This role is associated with an abundance of cervical mechanoreceptors. Recent studies have shown that proprioceptive training is associated with cervical joint position sense, joint range of motion, pain and disability. Also yoga combines physical exercises with breathing techniques and meditation and yoga is one of the most commonly used complementary treatments for neck pain.The aim of study is to determine the effectiveness of exercises for sensorimotor structure and yoga exercises with physical and meditative effects in individuals with chronic neck pain.

DETAILED DESCRIPTION:
Inclusion criteria for the study were: having a diagnosis of 'chronic neck pain', being over the age of 18, persistence of pain for more than 3 months, no neurogenic deficit, and agreeing to participate in the study. Exclusion criteria from the study are as follows: Having speech and comprehension problems, undergoing surgery on the neck region, having a history of trauma and cancer, and a diagnosis of vestibular disorder. After the analysis of the GPower 3.1 program to decide on the sample size, it was seen that a total of 50 participants should be included in the study for a statistical power of 82% (alpha:0.05). Participants diagnosed with chronic neck pain will be randomly divided into two groups as sensorimotor exercise group and yoga group by the evaluator. Sensorimotor exercise group; oculomotor exercise to provide information from the visual system, laser target exercise to provide information from the proprioception system, and postural stability exercise to provide information from the vestibular system. Yoga group will be given yoga exercises. Within the content of oculomotor exercise, gaze stability exercise and head-body coordination exercise will be given to the participants. Laser target exercise will be given with the laser target fixed on the participant's head and 90 cm away from the target. Postural stability exercise will be given in form of tandem exercise and standing on one leg. Yoga exercises will be applied by changing and combining 14 poses every week. The study will take 8 weeks. Participants in both groups will also be treated for 2 days a week. Participants will be evaluated twice, before and after treatment. Participants will be evaluated with Demographic Information Form, SF-36 Quality of Life Scale, Neck Disability Questionnaire, Tampa Kinesiophobia Scale, Numerical Pain Scale, Joint Range of Motion Measurement (G-Pro), Joint Position Error Test. Data analysis of the study will be done using SPSS 22.0 package program. The difference between Independent Groups will be compared with the Student's-t independent Test.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic neck pain at Grade 1 and 2 level,
* Being over 18 years old,
* Pain lasting more than 3 months,
* Absence of neurogenic deficit

Exclusion Criteria:

* Having been diagnosed with chronic neck pain at Grade 3 and 4 level,
* Having problems with speaking and understanding,
* Having undergone surgery on the neck region,
* Having a history of trauma,
* Having a history of cancer,
* Diagnosis of vestibular disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Short Form 36 Quality of Life Scale | Change in quality of life at 8 weeks
  SF-36 assesses quality of life by focusing on the physical, social and spiritual components of health. It consists of 36 items. Each item is scored between 0-100. 100 points indicate good health, 0 points poor health.
The Neck Disability Index | Change in functionality at 8 weeks
  The Neck Disability Index is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. Pain severity, personal care, concentration, driving, headache, lifting, working, sleeping, recretion, reading are questioned. This questionnaire consists of 10 questions, each question is given 0-5 points, and the higher the score, the higher the degree of disability. While 50 points is the highest possible score, 0 points is the lowest.
Tampa Kinesiophobia Scale | Change in fear of movement at 8 weeks
  Tampa Kinesiophobia Scale is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The questionnaire using 4 points to assess that are based on; the model of fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Numeric Pain Rating Scale | Change in pain intensity at 8 weeks
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults with chronic pain. NPRS is a segmented numeric version of the visual analog scale in which selects a whole number (0-10 integers) that best reflects the intensity of patients pain. An NPRS score of 3 and less than 3 represents low pain, 4-6 represents moderate pain, and greater than 7 represents severe pain.
Joint Range of Motion Measurement | Change in range of motion at 8 weeks
  Joint movements of the cervical region are performed using clinical instruments such as goniometer and cervical joint range of motion device. With the innovations brought by technology opportunities, different applications have been started to be used in the measurement of joint range of motion. The application named 'G-Pro' has good reliability and high validity in measuring active cervical joint range of motion in nonspecific neck pain participants. Participants will be evaluated with the G-Pro application. Values that should be in a healthy individual; 45-65 degrees for flexion, 45-50 degrees for extension, 55 degrees for rotation, and 40 degrees for lateral flexion.
Joint Position Error Test | Change in joint position sense at 8 weeks
  The Cervical Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. A target is placed on a wall 90cm away from the patient, at the patient's head height in sitting. The target is 90x80 cm in diameter. A laser pointer device is placed on the patient's head. The patient is then asked to focus on finding natural resting head position so that the laser pointer is in line with the centre. With eyes closed, the patient will actively move their head in one plane of motion and attempt to return to the starting position as accurately as possible. The patient should verbally indicate when they feel they have returned to the starting position. The distance of this point from the origin is measured. The more deteriorated the joint position sense is, the higher the value will be.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No